CLINICAL TRIAL: NCT03253172
Title: Renoprotective Effects of Potassium Supplementation in Chronic Kidney Disease (CKD)
Brief Title: Potassium Supplementation in CKD
Acronym: K+ in CKD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Dutch Kidney Foundation (Other); University Medical Center Groningen (Other); Leiden University Medical Center (Other); Amsterdam UMC (Other)
Responsible Party: Principal Investigator, Ewout Hoorn, Coordinating PI, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL60825.078.17; MEC-2017-226 (Other: ErasmusMC); CP16.01 (Other Grant/Funding Number: Dutch Kidney Foundation)
Record Dates: First submitted 2017-08-15; First posted 2017-08-17 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Renal Insufficiency, Chronic; Potassium Depletion; Hypertension; Hyperkalemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypokalemia; Hypertension; Hyperkalemia | interventions — Potassium Chloride; Potassium Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo
- Potassium Chloride (Experimental): Experimental Arm 1 - Rationale is that most evidence for a positive effect of potassium comes from studies using potassium chloride
  Interventions: Dietary Supplement: Potassium Chloride
- Potassium Citrate (Experimental): Experimental Arm 2 - Rationale for citrate is that recent evidence indicates that alkali treatment may also be renoprotective.
  Interventions: Dietary Supplement: Potassium Citrate

INTERVENTIONS:
Dietary Supplement: Potassium Chloride — Two potassium supplements with varying anions.
  Arms: Potassium Chloride
Dietary Supplement: Potassium Citrate — Potassium Citrate
  Arms: Potassium Citrate
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The current high-sodium, low-potassium diet contributes to the high prevalence of high blood pressure (hypertension). Indeed, the anti-hypertensive effects of potassium supplementation are well-established. Hypertension is even more prevalent and resistant in patients with chronic kidney disease (CKD) and contributes to further decline in kidney function. Four recent epidemiological studies (published 2014 - 2016) showed that higher dietary potassium intake was associated with better renal outcomes. All studies recommended an intervention study with potassium supplementation in patients with CKD, but this has not been performed. The aim of this study is to study the renoprotective effect of potassium supplementation in patients with CKD (stage 3b or 4, i.e. estimated glomerular filtration rate [eGFR] 15 - 45 ml/min/1.73 m2).

ELIGIBILITY:
Inclusion Criteria:

* CKD 3b or 4 (45 - 15 ml/min/1.73 m2)
* Δ eGFR (as estimated by the CKD-EPI equation) > 2 ml/min/1.73 m2/year (in preceding ≥ 1 year with at least 3 measurements)
* Hypertension (defined as office blood pressure > 140/90 mmHg or use of anti-hypertensive medication)

Exclusion Criteria:

* Hyperkalemia (serum potassium > 5.5 mmol/l) at study visit V0
* Medical reasons to continue dual RAAS-blockade, mineralocorticoid receptor blockers, potassium-sparing diuretics, or oral potassium binders.
* Patients with previous history of ventricular cardiac arrhythmia
* Patients with a life expectancy < 6 months
* Expected initiation of renal replacement therapy < 2 years
* Incapacitated subjects
* Women who are pregnant, breastfeeding or consider pregnancy in the coming 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Difference in estimated glomerular filtration rate (eGFR) | Two years

SECONDARY OUTCOMES:
≥ 30% decrease in eGFR | Two years
Slope analysis (change in eGFR in ml/min/1.73 m2/year) | Two years
Doubling in serum creatinine or end-stage renal disease | Two years
Progression to next CKD or albuminuria class | Two years
Ambulatory (24-hour) blood pressure | Two years
24-hour albuminuria | Two years
Cardiovascular event | Two years
  Coronary heart disease death, fatal myocardial infarction, fatal stroke and other cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, unstable angina, resuscitated cardiac arrest
All-cause mortality | Two years
Incidence of hyperkalemia | Two years
NT-pro-BNP | Two years
  Volume marker 1
Bioimpedance measures | Two years
  Volume marker 2
Pulse-wave velocity | Two years
  Cardiovascular marker 1
High-sensitive CRP | Two years
  Cardiovascular marker 2

OTHER OUTCOMES:
Effects of 2-week KCl supplementation on plasma potassium (mmol/l) | Two weeks
  Run-in outcome 1
Incidence of Hyperkalemia after 2-week KCl supplementation | Two weeks
  Run-in outcome 2
Effects of 2-week KCl supplementation on office blood pressure (mmHg) | Two weeks
  Run-in outcome 3

CONTACTS AND LOCATIONS:
Overall Officials: Ewout J Hoorn, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (4):
- Netherlands (4):
  - Academic Medical Center Amsterdam, Amsterdam
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sunga CGG, Zelnick LR, Bansal N. Urinary Sodium and Potassium Excretion and the Risk of Cardiovascular Events in CKD. Kidney360. 2026 Jan 1;7(1):94-106. doi: 10.34067/KID.0000000943. Epub 2025 Aug 8. No abstract available. PMID 40779318
- [Derived] Gritter M, Wouda RD, Yeung SMH, Wieers MLA, Geurts F, de Ridder MAJ, Ramakers CRB, Vogt L, de Borst MH, Rotmans JI, Hoorn EJ; on behalf of K onsortium. Effects of Short-Term Potassium Chloride Supplementation in Patients with CKD. J Am Soc Nephrol. 2022 Sep;33(9):1779-1789. doi: 10.1681/ASN.2022020147. Epub 2022 May 24. PMID 35609996